CLINICAL TRIAL: NCT07341490
Title: A Comparison of Computed Tomography-Angiography Versus Four-vessel Angiography in the Determination of Brain Death
Brief Title: CT-Angiography Versus Angiogram as Ancillary Tests in the Determination of Death by Neurologic Criteria
Acronym: Tadaa
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Peter Rudberg, M.D. Ph.D., Karolinska Institutet
Other Study IDs: 2025-4056
Record Dates: First submitted 2025-12-21; First posted 2026-01-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Infarction, Brain
Keywords: Cerebral infarction; Cerebral angiography; CT angiography; Brain Death; Diagnostic performance; Brain infarct
MeSH Terms: conditions — Brain Infarction; Cerebral Infarction; Brain Death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected Complete Cerebral Infarction: Patients with severe acute brain injury, in whom complete cerebral infarction has been declared by direct neurological criteria, but ancillary testing is warranted due to specific circumstances.

SUMMARY:
Diagnostic performance of a novel protocol for computed tomography-angiography, as ancillary test in the determination of complete cerebral infarction, in comparison to four vessel angiography.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Ongoing critical care due to severe acute brain injury
* Four vessel angiography necessary for the determination of complete cerebral infarction, according to Swedish legislation

Exclusion Criteria:

* Treatment with extracorporeal membrane oxygenation (ECMO)
* Radiologic examination by computed tomography deemed too challenging due to respiratory or circulatory instability, as determined by responsible clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving critical care
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance similar between computed tomography-angiography and four vessel angiography | Periprocedural
  Sensitivity, specificity, positive predictive value, negative predictive value, inter- and intrarater variability.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Observational, exploratory

DOCUMENTS (1):
  • Study Protocol (2025-11-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT07341490/Prot_000.pdf